CLINICAL TRIAL: NCT00634517
Title: A Multi-Center, Randomized, Double-Blind, Active-Controlled, Parallel Group, 4-Week Study to Evaluate the Efficacy, Safety and PK of Albuterol-HFA Versus Proventil-HFA in Pediatric Patients With Asthma in Pediatric Patients With Asthma
Brief Title: 4-Week Study of Efficacy, Safety and PK of Albuterol-HFA Versus Proventil-HFA in Pediatric Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IND voluntarily withdrawn, without prejudice
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-A004-CLN-E
Record Dates: First submitted 2008-03-07; First posted 2008-03-13 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T (Experimental): Armstrong Albuterol Sulfate Inhalation Aerosol, 216 mcg albuterol sulfate (108 mcg/actuation) is equivalent to 180 mcg albuterol base (90 mcg/actuation).
  Interventions: Drug: Armstrong Albuterol Sulfate Inhalation Aerosol
- R (Active Comparator): Proventil-HFA, Albuterol Sulfate Inhalation Aerosol, 216 mcg albuterol sulfate (108 mcg/actuation) is equivalent to 180 mcg albuterol base (90 mcg/actuation).
  Interventions: Drug: Albuterol Sulfate Inhalation Aerosol

INTERVENTIONS:
Drug: Armstrong Albuterol Sulfate Inhalation Aerosol — Albuterol Sulfate Inhalation Aerosol, 216 mcg albuterol sulfate (108 mcg/actuation) is equivalent to 180 mcg albuterol base (90 mcg/actuation).
  Other Names: Albuterol HFA
  Arms: T
Drug: Albuterol Sulfate Inhalation Aerosol — Albuterol Sulfate Inhalation Aerosol, 216 mcg albuterol sulfate (108 mcg/actuation) is equivalent to 180 mcg albuterol base (90 mcg/actuation).
  Other Names: Proventil-HFA
  Arms: R

SUMMARY:
This 4-week clinical study evaluates the efficacy and safety of Albuterol Sulfate HFA Inhalation Aerosol in comparison with the Active Control, Proventil-HFA (3M Pharmaceuticals, Inc) in pediatric patients (4-11 years old) with mild-to-moderate asthma. In addition, pharmacokinetic profile in this population will be evaluated using a population PK approach with sparse blood samples.

DETAILED DESCRIPTION:
This study consists of two periods:

1. Run-in Period (7-14 days): During the Run-in Period, subjects will maintain their current inhaled short-acting B2-agonist and inhaled corticosteroid therapies. All long-acting b-agonists (LABA) will be prohibited and replaced with a short-acting B2-agonist (Ventolin-HFA) and an inhaled corticosteroid, for a minimum of 7 days. Such LABA replacement therapy is not considered as violation of the asthma stability. The current orally inhaled corticosteroids may be maintained at the prescribed dosing regimen. All concomitant medications must be compliant or adjusted to the restrictions and washout time limits per Appendix II. Subjects will document their daily asthma symptom scores, treatment regimens, concomitant medications, PEF records, and adverse events if any.
2. Study Period (4 wk): During the 4-week Study Period, subjects will be randomized into one of the following 2 double-blinded treatment groups:

   * Treatment T (Albuterol-HFA, N=24): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), oral inhalation, QID;
   * Treatment R (Proventil-HFA, N=24): 216 mcg albuterol sulfate (equivalent to 180 mcg albuterol base), oral inhalation, QID.

During the Study Period, subjects will document their daily asthma symptom scores, treatment regimens, concomitant medications, PEF records, and adverse events if any. Three Clinical Visits are to be conducted, for measurement of treatment efficacy with serial spirometry (at Clinical Visit 1 and 3); for monitoring safety and compliance (at Clinical Visit 1, 2 and 3); and for evaluating pharmacokinetic profiles in part of the study population (greater than or equal to 6 subjects per Arm) using a population PK approach (PPK) with a sparse blood sampling regimen (at Clinical Visit 3).

STUDY POPULATION

Sufficient enrollment will be planned to obtain 48 subjects as "Per protocol population", with 24 in Albuterol-HFA (Arm T) and 24 in the Proventil-HFA (Arm R). Qualified subjects should be:

1. Male and female patients aged 4 - 11 years (upon screening), and female patients being premenarchal upon Visit-1.
2. With documented mild-to-moderate asthma for at least 6 months prior to screening;
3. Being able to reliably perform spirometric FEV1 test;
4. Consent, under supervision of a parent or a legal guardian, to participate in the study;
5. Having a baseline forced expiratory volume in 1 second (FEV1) that is 50.0%-100.0% of predicted values at screening (Screening Baseline FEV1);
6. Demonstrating a greater than or equal to 12.0% FEV1 reversibility in the Reversibility Test, at 30 min after inhaling 180 mcg of Ventolin-HFA;
7. Satisfying the criterion of asthma stability, defined as no significant changes in asthma therapy and no asthma-related hospitalization or emergency visits, over 4 weeks prior to the screening;
8. Satisfying the Run-in Period requirements;
9. Satisfying all other inclusion/exclusion criteria, as specified in Section 4.2.

TREATMENT REGIMENS

Enrolled subjects will be randomized to receive one of the 2 double-blinded treatments: Albuterol-HFA (Treatment T) or Proventil-HFA (Treatment R).

CLINICAL VISITS:

The entire study consists of a Screening Period, a Run-in Period, and a Study Period which consists of three (3) Clinical Visits. The three (3) Clinical Visits are scheduled with 14±3 days intervals, as Visit 1 (Day 0 of treatment), Visit 2 (Day 14), and Visit 3 (Day 28). The Clinical Visit 1 will be held within 7-14 days after Screening Visit. Serial FEV1 are performed at Visit 1 and 3. Safety and compliance are evaluated at all 3 Visits. Population PK (PPK) blood sampling is conducted at Visit 3.

METHODOLOGIES AND SPECIFIC MEASUREMENTS

1. Forced Expiratory Volume at 1st Second (FEV1)

   Spirometry is to be used to determine Forced Expiratory Volume in the 1st second (FEV1). Patient may choose either a standing or a sitting position for FEV1. The position, once chosen, should be kept consistent for the entire study. Nose clips will be worn for the FEV1 measurements.

   Each FEV1 is measured in triplicate at a given test or a given time point. The highest FEV1 volume, from the triplicate attempts, is used as the representative value. The highest and second highest FEV1 attempts should not differ by greater than 0.2 L. Up to 2 additional attempts may be measured if necessary, with a total of 3-5 attempts allowed for a given test. The accepted attempts have to be technically conforming to the current spirometry standards from the American Thoracic Society (ATS). The current clinical normative lung volumes in conformity with the ATS guidelines will be used for calculating the predicted percentage.
2. Peak Expiratory Flow (PEF) Rate

PEF will be measured as a means of monitoring safety and asthma control. PEF will be measured in triplicate, with additional attempts if necessary. The highest PEF volume is used as the representative value. Two measurements of PEF are made daily, once prior to the first AM dose and once prior to the last PM dose of the study drug. Subject will be standing for PEF measurements. No nose-clips will be needed for PEF.

2) Screening Baseline FEV1

Passing the Screening Baseline FEV1 test is one of the prerequisites for enrollment, and is to be conducted at the Screening Visit by all subjects. The Screening Baseline FEV1 should fall within 50.0%-100.0% of the predicted value to qualify the subject.

3) Reversibility FEV1 Test

Reversibility FEV1 Test will be performed at the Screening Visit. Within 30 min after the Screening Baseline FEV1 is obtained, the subject will self-administer 180 to 360 mcg Ventolin-HFA (2-4 inhalations). To qualify for the study, the subject needs to demonstrate an FEV1 reversibility of greater than or equal to 12.0%, from the (same-day) Screening Baseline FEV1, with 3 to 8 attempts, at 30 min after inhaling Ventolin-HFA. Reversibility is defined as:

% Reversibility = [(FEV1 postdose ~ FEV1 predose)/FEV1 predose] x 100%

Up to two-time re-tests of the Reversibility FEV1 Test will be allowed if the highest attempted reversibility value is less than 12.0% but greater than or equal to 6.0, if deemed necessary by the investigator, with screening period extendable to a total of 21 days.

4) Serial FEV1 measurements of study drug efficacy

Response to the study drugs (T and R) is examined by serial spirometric measurements of FEV1 post-dose. Serial FEV1 will be conducted at each of the following time points during Study Visits 1 and 3:

1. at baseline (within 30 minutes prior to study drug dosing).
2. at 10, 30, 45, 60, 120, 180, 240, 300, and 360 minutes after dosing.

POPULATION PHARMACOKINETIC (PPK) EVALUATION

At clinical Visit 3, a sufficient number of patients will be subject to a population pharmacokinetic (PPK) study to obtain a minimum of 6 subjects per arm with complete and correct 4 PK samples. An indwelling IV catheter may be used, as an alternative to repeated venipunctures, for PPK samples. An appropriate anticoagulant may be used to maintain the catheter patency. Four blood samples (~5.0 mL each) will be taken from a hand or forearm vein of the subject, at pre-scheduled 4 time points: 2, 4, 6 and 8 hr post-dose (each with a ±15 min window). No inhalation of the study drug or rescue medication should take place until completion of the 8-hr PK sampling, unless needed for rescue, at which point the subject will not be considered evaluable for the PK endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy.
2. Male and female mild-to-moderate asthma patients.
3. Aged 4 - 11 yr (upon screening).
4. Female patients must be premenarchal upon Visit-1, and those who become menarchal during the study must use an accepted method of contraception including abstinence.
5. A documented history of asthma, for at-least 6-months prior to Screening, requiring inhaled B-adrenergic agonists, with or without inhaled corticosteroids for asthma symptom control.
6. Satisfying asthma stability criterion, defined as no changes in asthma therapy and no asthma-related hospitalization or emergency room visits, over the 4 weeks prior to Screening.
7. Being able to withhold treatment with inhaled bronchodilators and/or restricted medications for the minimum washout periods indicated in Appendix II, for the purpose of conducting clinical visits.
8. Having a baseline forced expiratory volume in 1 second (FEV1), that is 50.0-100.0% of predicted values at the screening (Screening Baseline FEV1).
9. Demonstrating a greater than or equal to 12.0% reversibility in the Reversibility Test, at 30 min after inhaling 2-4 puffs (180-360 mcg) of Ventolin-HFA.
10. Demonstrating correct use of metered-dose inhaler (MDIs), and acceptable performance in the FEV1 measurements.
11. Has properly consented, with a parent or a legal guardian, to participate in this study.

Exclusion Criteria:

1. Any current or past significant medical conditions that, according to the investigator, might affect pharmacodynamic response to the study drugs, such as significant systemic or respiratory diseases (e.g., cystic fibrosis, bronchiectasis, emphysema, nonreversible pulmonary diseases), other than asthma.
2. Concurrent clinically significant cardiovascular, hematological, renal, neurological, hepatic, and endocrine disorders, or psychiatric diseases.
3. Known intolerance or hypersensitivity to any component of the MDI formulation (e.g., albuterol, HFA-134a, oleic acid, ethanol).
4. Recent upper (within 2 weeks) or lower (within 4 weeks) respiratory tract infection before screening.
5. Recent (within 4 weeks) use of systemic (or oral) corticosteroids and B-adrenergic bronchodilators; or recent (within 2 weeks) use of monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), or B-blockers; before the Screening.
6. Having been on other investigational drug/device studies in the last 30 days prior to screening.
7. Known or reasonably suspected alcohol/drug abuses.
8. Having smoked within the last 12 months.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for efficacy evaluation is to obtain the ratio of the geometric mean of area under the curve of change in FEV1%versus time for pediatric patients using the study drug to the active reference drug. | visits 1 and 3

SECONDARY OUTCOMES:
AUC of serial FEV1 volume changes from the Same Day Baseline versus time, during the 6-hr post-dose. | each visit
Time to onset of bronchodilator effect, determined by linear interpolation as the time point when FEV1 first exceeded 12.0% over the respective Same Day Baseline. | each visist
The peak bronchodilator response, Fmax, defined as the maximum FEV1 (% change from the Same Day Baseline). | each visit
The time to peak bronchodilator response (FEV1), with Fmax defined as the maximum FEV1 (% change from the Same Day Baseline). | each visit
Duration of bronchodilator effect, defined as the total duration when FEV1 is maintained greater than or equal to 12.0% above the respective Same Day Baseline values. | each visit
(6) Percentage of positive responders including those whose FEV1 exceed the Same-Day Baseline by greater than or equal to 12.0% at or before 30 min post-dose (quick responders), and at any time during the entire 6 hr post-dose (overall responders). | each visit
Pharmacokinetic parameters including Cmax, AUC, and t1/2, based on a population pharmacokinetic (PPK) approach with sparse blood samples, conducted at Clinical Visit 3. | visit 3
Requirements for rescue/concomitant medications, for each treatment group | end of study
Mean Overall Asthma Control Scores evaluated by investigators | end of study
Total daytime asthma symptom scores | end of study
Nighttime sleep disturbance scores | end of study
Morning and evening pre-dose Peak Expiratory Flow Rate (PEF). | end of study
Number of asthma exacerbations during the entire study period | end of study
Vital signs (SBP/DBP, and heart rate) will be monitored at: 1. baseline (prior to dosing), and; 2. 60 minutes post-dose, but before the 60 min FEV1 tests. 3. 360 minutes post-dose, but before the 360 min FEV1 tests. | Screening, visits 1 and 3
A 12-lead ECG (HR, QT and QTc intervals) recorded at: 1. pre-dose, and; 2. 60 minutes post-dose, but before the 60 min FEV1 tests. | Screening and visits 1 and 3
lab tests for CBC, blood metabolic panel, and urinalysis. | Pre-study and end of study
Physical examinations | Screening and end of study
Blood potassium levels | Screening and EOS for all subjects; and at 120+15 min post dose (Visit 3) for population PK subjects only
Study compliance and safety will be reviewed. Concomitant medications will be reviewed and recorded | All Study Visits
Adverse events, whether observed by investigators or reported by subjects, will be documented and followed up if deemed necessary. | At All Study Visits

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - West Coast Clinical Trials Phase 2-4, LLC, Long Beach, California
  - Allergy Associates Medical Group, Inc., San Diego, California
  - Bensch Research Associates, Stockton, California
  - Integrated Medical Research, Ashland, Oregon
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas